CLINICAL TRIAL: NCT01855789
Title: A Randomized, Double-Blind Trial Assessing the Impact of Methotrexate Discontinuation on the Efficacy of Subcutaneous Tocilizumab With Methotrexate Therapy
Brief Title: A Study of the Impact of Methotrexate (MTX) Discontinuation on the Efficacy of Subcutaneous (SC) Tocilizumab (TCZ) With MTX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML28776
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Non-Randomized Participants (TCZ + MTX) (Experimental): All participants will receive initial treatment with open-label TCZ + MTX. Participants who complete 24-week treatment with open-label TCZ + MTX and did not achieve a DAS28 score </=3.2 at Week 24, will continue receiving TCZ + MTX in open label manner up to Week 52.
  Interventions: Drug: Tocilizumab (TCZ); Drug: Methotrexate (MTX)
- Randomized Participants (TCZ + MTX) (Experimental): Participants who complete the initial 24-week treatment with open-label TCZ + MTX and achieve a DAS28 score </=3.2 at Week 24, will be randomized to receive TCZ along with MTX up to Week 52.
  Interventions: Drug: Tocilizumab (TCZ); Drug: Methotrexate (MTX)
- Randomized Participants (TCZ + PBO) (Active Comparator): Participants who complete the initial 24-week treatment with open-label TCZ + MTX and achieve a DAS28 score </=3.2 at Week 24, will be randomized to receive TCZ along with MTX matched placebo (PBO) up to Week 52.
  Interventions: Drug: Tocilizumab (TCZ); Drug: Placebo (PBO)

INTERVENTIONS:
Drug: Tocilizumab (TCZ) — TCZ will be administered at a dose of 162 milligrams (mg) via SC injection weekly (if body weight is greater than or equal to [>/=] 100 kilograms [kg]) or every 2 weeks (if body weight was less than [<] 100 kg).
  Other Names: Actemra
Drug: Methotrexate (MTX) — MTX will be administered at a stable dose (15 mg to 25 mg per week) orally.
  Arms: Non-Randomized Participants (TCZ + MTX); Randomized Participants (TCZ + MTX)
Drug: Placebo (PBO) — PBO matching to MTX will be administered orally.
  Arms: Randomized Participants (TCZ + PBO)

SUMMARY:
This randomized, multicenter, double-blind, parallel group study will evaluate the impact of MTX discontinuation on the efficacy of SC TCZ in participants with moderate to severe active rheumatoid arthritis who have an inadequate response to current MTX therapy. Participants will initiate treatment with TCZ weekly or every 2 weeks along with MTX at a stable dose orally in an open-label manner for 24 weeks. Participants with a disease activity score based on 28 joints (DAS28) less than or equal to (</=) 3.2 at Week 24, will be randomized to either continue receiving a stable dose of MTX or to switch to matching placebo up to Week 52. Participants without a DAS28 score </=3.2 at Week 24, will continue the same treatment in a non-randomized open-label manner up to Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Body weight </=150 kg
* Active moderate to severe rheumatoid arthritis (DAS28 >/=4.4) according to the revised 1987 ACR criteria at screening and baseline (prior to treatment on Day 1)
* Currently receiving oral MTX for at least 24 weeks and on a stable oral dose of at least 15 mg/week for at least 6 weeks prior to treatment (Day 1), with the following exception: a stable dose of at least 10 mg/week is allowed for participants with a body weight <50 kg or calculated glomerular filtration rate (or creatinine clearance) <60 milliliters per minute (mL/min)
* History of parenteral (SC or intramuscular [IM]) MTX is allowed, but not within 6 weeks prior to treatment (Day 1). Participants must not have a documented, clinically significant intolerance to oral MTX and must be receiving oral MTX at a dose of 15 mg/week for at least 6 weeks prior to treatment (Day 1)
* Participants who have received one prior anti-tumor necrosis factor (TNF) must have discontinued etanercept, infliximab, certolizumab, adalimumab, or golimumab for at least 6 months prior to screening
* Oral corticosteroids must have been </=10 mg/day prednisone (or equivalent) and stable for at least 25 out of 28 days prior to treatment (Day 1)
* Participants receiving treatment on an outpatient basis

Exclusion Criteria:

* Documented medical history of significant intolerance to oral MTX >/=15 mg/week
* Participants receiving other (non-MTX) disease modifying anti-rheumatic drugs (DMARDs) within 8 weeks of screening
* Previous treatment with abatacept, rituximab, tofacitinib, or anakinra
* Treatment with parenteral corticosteroids within 4 weeks prior to treatment
* Previous treatment with cell-depleting therapies or alkylating agents
* Previous treatment with TCZ
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery during the study
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Non-rheumatic active autoimmune diseases (for example, inflammatory bowel diseases, psoriasis, multiple sclerosis)
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* Functional Class IV according to the revised (1987) ACR criteria for rheumatoid arthritis
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of significant uncontrolled concomitant diseases; uncontrolled disease states where flares are commonly treated with oral or parenteral corticosteroids
* Active current or history of recurrent infection, or any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks prior to screening or oral antibiotics within 2 weeks prior to screening
* Active tuberculosis requiring treatment within the previous 3 years
* History of or currently active primary or secondary immunodeficiency
* Pregnant or breast-feeding women
* Positive for hepatitis B or hepatitis C infection
* For potential MRI substudy participants: the presence of any metal-containing device or object in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (155):
- United States (155):
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Uni Of Alabama,Birmingham; Medicine - Rheumatology, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Clnical & Translational Reseach Center for Alabama, PC, Tuscaloosa, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, Pllc, Mesa, Arizona
  - Arizona Arthritis and Rheuma, Mesa, Arizona
  - Valley Arthritis Care, Phoenix, Arizona
  - Advanced Arthritis Care & Research, Scottsdale, Arizona
  - Fort Smith Rheumatology, PC, Fort Smith, Arkansas
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph, Fullerton, California
  - CV Mehta MD Medical Corp, Hemet, California
  - Valerius Medical Group, Los Alamitos, California
  - NRC Research Institute, Orange, California
  - San Diego Arthritis Med Clnc, San Diego, California
  - C Michael Neuwelt MD Inc, San Leandro, California
  - Inland Rheumatology; Clinical Trials, Inc., Upland, California
  - Medvin Clinical Research, Whittier, California
  - University of Colorado Hospital, Aurora, Colorado
  - Arthritis Assoc & Osteoporosis; Ctr of Colorado Springs, Colorado Springs, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Joao Nascimento, Bridgeport, Connecticut
  - Clinical Research Center of Ct/Ny, Danbury, Connecticut
  - Arthritis & Osteoporosis Center Pc, Hamden, Connecticut
  - New England Research Associates, Trumbull, Connecticut
  - Rheumatolgy Consultants of Deleware, Lewes, Delaware
  - Javed Rheumatology Associates, Inc., Newark, Delaware
  - Arthritis & Rheumatism; Disease Specialities, Aventura, Florida
  - Robert Levin, Md; Research Dept, Dunedin, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - South Coast Research Center, Inc., Miami, Florida
  - Precision Research Organization, Miami Lakes, Florida
  - Jeffrey Alper M.D Research, Naples, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Arthritis and Rheumatology Clinic, Orlando, Florida
  - Arthritis Center Palm Harbor, Palm Harbor, Florida
  - Arthritis Rsrch of Florida, Inc., Palm Harbor, Florida
  - Sarasota Arthritis Res Center, Sarasota, Florida
  - Pinellas Medical Research - Allegry & Rheumatology Associates, LLC, St. Petersburg, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - McIlwain Medical Group, Tampa, Florida
  - Burnette & Silverfield, MDS, Tampa, Florida
  - Advanced Clinical Research of Orlando, Inc., Winter Garden, Florida
  - North Georgia Rheumatology, Duluth, Georgia
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - North Georgia Rheumatology Group, PC, Lawrenceville, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Springfield Clinic, Springfield, Illinois
  - Indiana Uni Medical Center, Indianapolis, Indiana
  - Diagnostic Rheumatology & Research, Indianapolis, Indiana
  - Kansas City Internal Medicine, Overland Park, Kansas
  - Bluegrass Comm Research, Inc., Lexington, Kentucky
  - Arthritis & Diabetes Clinic, Inc, Monroe, Louisiana
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - New England Medical Center; Dept. of Medicine, Div. of Rheumatology, Boston, Massachusetts
  - Phase Iii Clinical Research, Fall River, Massachusetts
  - Mansfield Medical Center, Mansfield, Massachusetts
  - Reliant Medical Group, Inc; Rheumatology, Worcester, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Advanced Rheumatology, PC, Lansing, Michigan
  - Fiechtner Research Inc, Lansing, Michigan
  - Nisus Research/Northern Michigan Hospital, Petoskey, Michigan
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - St. Luke's Hospital Association of Duluth, Duluth, Minnesota
  - St. Paul Rheumatology, Eagan, Minnesota
  - Arthritis and Osteoporosis; Treatment and Research Center, Flowood, Mississippi
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - David S Rosenberg, Florissant, Missouri
  - Clinical Research Consultants,LLC, Kansas City, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Arthritis Consultants, St Louis, Missouri
  - G. T. Kelly, MD, Las Vegas, Nevada
  - Rheumatology Research Group, Lebanon, New Hampshire
  - Nashua Rheumatology - Foundation Medical Partners, Nashua, New Hampshire
  - Arthritis and Osteoporosis Associates, Manalapan, New Jersey
  - Atlantic Coast Rheumatology, Toms River, New Jersey
  - Ocean Rheumatology, Toms River, New Jersey
  - Arthritis Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - The Center for Rheumatology, Albany, New York
  - Arthritis & Osteoporosis Center, Brooklyn, New York
  - Manhasset Rheumatology, Manhasset, New York
  - Manhattan Medical Reserach, New York, New York
  - Buffalo Rheumatology Associates, Orchard Park, New York
  - Office of Premier Chatpar Md, Plainview, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Arthritis Health Associates, Syracuse, New York
  - Asheville Arthritis & Osteoporosis Center, PA, Asheville, North Carolina
  - Carolina Bone & Joint P.A., Charlotte, North Carolina
  - Triangle Orthopaedics Associates, P.A., Durham, North Carolina
  - Medication Management, Greensboro, North Carolina
  - PMG Research of Hickory LLC, Hickory, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Shanahan Rheumatology & Immunology, PLLC, Raleigh, North Carolina
  - St. Alexius Medical Center; Arthritis Clinic, Bismarck, North Dakota
  - Odyssey Research Services; Main Medical Building, Bismarck, North Dakota
  - Crystal Arthritis Center, Inc., Akron, Ohio
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University; Rheumatology; Immun/Rheum, Columbus, Ohio
  - Columbus Arthritis Center, Columbus, Ohio
  - STAT Research Inc, Dayton, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Clinical Research Source, Inc., Toledo, Ohio
  - Arthritis Care Center Oklahoma, Ardmore, Oklahoma
  - Arthritis and Rheumatology; Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - Health Research of Oklahoma, Llc, Oklahoma City, Oklahoma
  - Lynn Health Science Inst., Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Arthritis Associates, Erie, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, Wexford, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Emkey Arthritis & Osteoporosis, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Columbia Arthritis Center (Partnership Practice), Columbia, South Carolina
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh Gupta - PP, Memphis, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Lovelace Scientific Resources Inc., Austin, Texas
  - Diagnostic Group, Beaumont, Texas
  - AOCBV, College Station, Texas
  - Adriana Pop-Moody MD Clinic PA, Corpus Christi, Texas
  - Arthritis Care & Diagnostic Center, Dallas, Texas
  - Metroplex Clinical Research, Dallas, Texas
  - Rheumatic Disease Clin Res Ctr, Houston, Texas
  - IntraFusion Researh Network, Houston, Texas
  - Houston Inst. For Clinical Research, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - Accurate Clinical Management, San Antonio, Texas
  - NextGen Clinical Research Inc, San Antonio, Texas
  - Arthiritis & Osteoporosis Centre of South Texas, San Antonio, Texas
  - Arthritis Clinic Of Central Texas, San Marcos, Texas
  - Crossroads Clinical Research, LLC, Victoria, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
  - South Puget Sound Clinical Research, Olympia, Washington
  - Arthritis Northwest, Spokane, Spokane, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Rheumatic Disease Center, Glendale, Wisconsin
  - Lakeshore Orthopedics, Manitowoc, Wisconsin
  - Gundersen Clinic Ltd;Sec. Rheumatology/Dept. of Internal Med, Onalaska, Wisconsin

REFERENCES:
- [Derived] Kremer JM, Rigby W, Singer NG, Birchwood C, Gill D, Reiss W, Pei J, Michalska M. Sustained Response Following Discontinuation of Methotrexate in Patients With Rheumatoid Arthritis Treated With Subcutaneous Tocilizumab: Results From a Randomized, Controlled Trial. Arthritis Rheumatol. 2018 Aug;70(8):1200-1208. doi: 10.1002/art.40493. Epub 2018 Jun 14. PMID 29575803

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized participants constituted the primary analysis population for the efficacy assessments, while all other analyses including safety assessments were performed on overall study population. An MRI sub-study was planned to evaluate joint inflammation in conjunction with other clinical signs and symptoms.
Groups:
- Period 1: All Participants (TCZ + MTX): All enrolled participants received tocilizumab (TCZ) at a dose of 162 milligrams (mg) via subcutaneous (SC) injection weekly (qw; if body weight was greater than or equal to [>/=] 100 kilograms [kg]) or every 2 weeks (q2w; if body weight was less than [<] 100 kg) along with methotrexate (MTX) at a stable dose (15 mg to 25 mg per week) in an open-label manner orally for 24 weeks. Participants, who achieved a disease activity score based on 28 joints (DAS28) less than or equal to (</=) 3.2 at Week 24, were randomized and received double-blind treatment according to the arm in which they were randomized (TCZ + MTX or TCZ + PBO [placebo]) up to Week 52. Participants who did not achieve a DAS28 score </=3.2 at Week 24 continued the same treatment in a non-randomized open-label manner up to Week 52.
- Period 2: Randomized Participants (TCZ + MTX): Participants, who completed the initial 24-week treatment with TCZ + MTX and achieved a DAS28 score </=3.2 at Week 24, were randomized and received TCZ at a dose of 162 mg via SC injection qw or q2w along with MTX at a stable dose orally up to Week 52.
- Period 2: Randomized Participants (TCZ + PBO): Participants, who completed the initial 24-week treatment with TCZ + MTX and achieved a DAS28 score </=3.2 at Week 24, were randomized and received TCZ at a dose of 162 mg via SC injection qw or q2w along with MTX matched placebo (PBO) orally up to Week 52.
- Period 2: Non-Randomized Participants (TCZ + MTX): Participants, who completed the initial 24-week treatment with TCZ + MTX and did not achieve a DAS28 score </=3.2 at Week 24, continued receiving TCZ at a dose of 162 mg via SC injection qw along with MTX in open label manner orally up to Week 52.
Period: 1) Baseline up to Week 24
Arm/Group | Period 1: All Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO) | Period 2: Non-Randomized Participants (TCZ + MTX)
Started | 718 | 0 | 0 | 0
Completed | 602 | 0 | 0 | 0
Not Completed | 116 | 0 | 0 | 0
Not completed — Adverse Event | 37 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 16 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 31 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Participant Non-compliance | 3 | 0 | 0 | 0
Not completed — Sponsor Decision | 3 | 0 | 0 | 0
Not completed — Other | 4 | 0 | 0 | 0
Period: 2) Week 24 up to End of Study
Arm/Group | Period 1: All Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO) | Period 2: Non-Randomized Participants (TCZ + MTX)
Started | 0 | 147 | 147 | 308
Completed | 0 | 132 | 129 | 250
Not Completed | 0 | 15 | 18 | 58
Not completed — Adverse Event | 0 | 4 | 5 | 21
Not completed — Serious Hypersensitivity Reaction | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 5 | 16
Not completed — Lost to Follow-up | 0 | 1 | 1 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 7 | 5 | 8
Not completed — Physician Decision | 0 | 0 | 2 | 4
Not completed — Participant Non-compliance | 0 | 1 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy assessment.
Groups:
- Overall Study Population: All enrolled participants received TCZ at a dose of 162 mg via SC injection qw (if body weight was >/=100 kg) or q2w (if body weight was <100 kg) along with MTX at a stable dose (15 mg to 25 mg per week) in an open-label manner orally for 24 weeks. Participants, who achieved a DAS28 score </=3.2 at Week 24, were randomized and received double-blind treatment according to the arm in which they were randomized (TCZ + MTX or TCZ + PBO) up to Week 52. Participants who did not achieve a DAS28 score </=3.2 at Week 24 continued the same treatment in a non-randomized open-label manner up to Week 52.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 556
  Male | 155

OUTCOME MEASURES:

1. Primary Outcome: Change From Week 24 in Disease Activity Score Based on 28 Joints (DAS28) Score at Week 40
Description: The DAS28 was derived from assessments of erythrocyte sedimentation rate (ESR) measured in millimeters per hour (mm/h), tender joint count on 28 joints (TJC28), swollen joint count on 28 joints (SJC28), and Patient's Global Assessment of disease activity according to 100--millimeter (mm) Visual Analog Scale (VAS). DAS28 score was calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28 score could range from 0 to 10, where higher score represented higher disease activity. The change from Week 24 to Week 40 was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Week 24, Week 40
Population: Analysis was performed on randomized group which included participants in ITT population who were randomized and received blinded treatment at Week 24. Missing Week 40 values were imputed using last available assessment obtained after Week 24. Here, 'Number Analyzed' signifies number of participants with assessment at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
units on a scale
  Week 24 | 2.13 (0.816) | 2.11 (0.822)
  Change at Week 40: number analyzed (Participants) | 146 | 147
  Change at Week 40 | 0.15 (1.127) | 0.48 (1.275)
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Analysis of covariance (ANCOVA) model included Week 24 DAS28 as a covariate, treatment group, and the randomization stratification factors: DAS28 remission status at Week 24 (<2.6, >/=2.6 to </=3.2), baseline weight-by-dosing group (<80 kg q2w, <80 kg qw, 80-<100 kg q2w, 80-<100 kg qw, >/=100 kg qw), participant anti-tumor necrosis factor (anti-TNF) exposure (Yes/No); Test type: Non-Inferiority — Non-inferiority of TCZ + PBO was claimed if the upper bound of the 95% confidence interval (CI) for the mean difference was below 0.6; Estimated Mean Difference = 0.318, 95% CI 2-sided [0.045 to 0.592], Standard Error of Mean 0.139

2. Secondary Outcome: Percentage of Participants Achieving 20% Improvement in American College of Rheumatology (ACR20) Response
Description: The ACR20 response at any time was defined as >/=20% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 20% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) Patient's global assessment of disease activity according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via a Health Assessment Questionnaire-Disability Index (HAQ-DI), and 5) Acute phase reactant (ESR in mm/h or C-Reactive Protein [CRP] in milligrams per deciliter [mg/dL]).
Time Frame: Weeks 24, 40, and 52
Population: Analysis was performed on randomized group. Missing assessments of response were treated as no response.
Measure: Number; unit: percentage of participants
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
percentage of participants
  Week 24 | 91.2 (0.816) | 83.0 (0.822)
  Week 40 | 78.9 (1.127) | 68.7 (1.275)
  Week 52 | 74.1 | 65.3
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 40: Analysis of association between treatment group and response, stratified by the randomization stratification factors: DAS28 remission status at Week 24 (<2.6, >=2.6 to <=3.2), baseline weight-by-dosing group (<80 kg q2w, <80 kg qw, 80-<100 kg q2w, 80-<100 kg qw, >=100 kg qw), participant anti-TNF exposure (Yes/No); Test type: Superiority; p = 0.0746, Cochran-Mantel-Haenszel; ACR 20 Response Rate Difference = -10.2, 95% CI 2-sided [-20.2 to -0.2] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented
Statistical Analysis 2: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 52: Analysis of association between treatment group and response, stratified by the randomization stratification factors: DAS28 remission status at Week 24 (<2.6, >=2.6 to <=3.2), baseline weight-by-dosing group (<80 kg q2w, <80 kg qw, 80-<100 kg q2w, 80-<100 kg qw, >=100 kg qw), participant anti-TNF exposure (Yes/No); Test type: Superiority; p = 0.1159, Cochran-Mantel-Haenszel; ACR 20 Response Rate Difference = -8.8, 95% CI 2-sided [-19.3 to 1.6] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented
Statistical Analysis 3: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 24; Test type: Superiority; ACR 20 Response Rate Difference = -8.2, 95% CI 2-sided [-15.8 to -0.6] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented

3. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in American College of Rheumatology (ACR50) Response
Description: The ACR50 response at any time was defined as >/=50% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 50% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) Patient's global assessment of disease activity according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via HAQ-DI, and 5) Acute phase reactant (ESR in mm/h or CRP in mg/dL).
Time Frame: Weeks 24, 40, and 52
Population: Analysis was performed on randomized group. Missing assessments of response were treated as no response.
Measure: Number; unit: percentage of participants
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
percentage of participants
  Week 24 | 74.1 (0.816) | 63.3 (0.822)
  Week 40 | 63.9 (1.127) | 50.3 (1.275)
  Week 52 | 62.6 | 47.6
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0377, Cochran-Mantel-Haenszel; ACR 50 Response Rate Difference = -13.6, 95% CI 2-sided [-24.8 to -2.4] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented
Statistical Analysis 2: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0130, Cochran-Mantel-Haenszel; ACR 50 Response Rate Difference = -15.0, 95% CI 2-sided [-26.2 to -3.7] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented
Statistical Analysis 3: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 24; Test type: Superiority; ACR 50 Response Rate Difference = -10.9, 95% CI 2-sided [-21.4 to -0.4] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented

4. Secondary Outcome: Percentage of Participants Achieving 70% Improvement in American College of Rheumatology (ACR70) Response
Description: The ACR70 response at any time was defined as >/=70% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 70% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) Patient's global assessment of disease activity according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via HAQ-DI, and 5) Acute phase reactant (ESR in mm/h or CRP in mg/dL).
Time Frame: Weeks 24, 40, and 52
Population: Analysis was performed on randomized group. Missing assessments of response were treated as no response.
Measure: Number; unit: percentage of participants
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
percentage of participants
  Week 24 | 45.6 (0.816) | 37.4 (0.822)
  Week 40 | 42.2 (1.127) | 34.0 (1.275)
  Week 52 | 48.3 | 36.7
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3599, Cochran-Mantel-Haenszel; ACR 70 Response Rate Difference = -8.2, 95% CI 2-sided [-19.2 to 2.9] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented
Statistical Analysis 2: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0663, Cochran-Mantel-Haenszel; ACR 70 Response Rate Difference = -11.6, 95% CI 2-sided [-22.8 to -0.3] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented
Statistical Analysis 3: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 24; Test type: Superiority; ACR 70 Response Rate Difference = -8.2, 95% CI 2-sided [-19.4 to 3.1] — Observed difference in percentages (TCZ + PBO minus TCZ + MTX) and the asymptotic Wald 95% CI is presented

5. Secondary Outcome: Percentage of Participants With >/=1.2 Points Increase (Worsening) From Week 24 in DAS28 Score at Week 40 and 52
Description: The DAS28 was derived from assessments of ESR measured in mm/h, TJC28, SJC28, and Patient's global assessment of disease activity according to 100-mm VAS. DAS28 score was calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28- score could range from 0 to 10, where higher score represented higher disease activity.
Time Frame: Week 24, 40, and 52
Population: Analysis was performed on randomized group. Missing assessments of DAS28 were treated as worsening.
Measure: Number; unit: percentage of participants
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
percentage of participants
  Week 40 | 21.1 (0.816) | 28.6 (0.822)
  Week 52 | 26.5 (1.127) | 29.9 (1.275)
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 40: Analysis of association between treatment group and worsening in DAS28, stratified by the randomization stratification factors: DAS28 remission status at Week 24 (<2.6, >=2.6 to <=3.2), baseline weight-by-dosing group (<80 kg q2w, <80 kg qw, 80-<100 kg q2w, 80-<100 kg qw, >=100 kg qw), participant anti-TNF exposure (Yes/No); Test type: Superiority; p = 0.2371, Cochran-Mantel-Haenszel; DAS28 Worsening Rate Difference = 7.5, 95% CI 2-sided [-2.4 to 17.3] — TCZ + PBO minus TCZ + MTX
Statistical Analysis 2: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); Week 52: Analysis of association between treatment group and worsening in DAS28, stratified by the randomization stratification factors: DAS28 remission status at Week 24 (<2.6, >=2.6 to <=3.2), baseline weight-by-dosing group (<80 kg q2w, <80 kg qw, 80-<100 kg q2w, 80-<100 kg qw, >=100 kg qw), participant anti-TNF exposure (Yes/No); Test type: Superiority; p = 0.4811, Cochran-Mantel-Haenszel; DAS28 Worsening Rate Difference = 3.4, 95% CI 2-sided [-6.9 to 13.7] — TCZ + PBO minus TCZ + MTX

6. Secondary Outcome: Percentage of Participants With DAS28 Score <2.6 (DAS28 Remission)
Description: The DAS28 was derived from assessments of ESR measured in mm/h, TJC28, SJC28, and Patient's global assessment of disease activity according to 100-mm VAS. DAS28 score was calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28 score could range from 0 to 10, where higher score represented higher disease activity.
Time Frame: Week 40, Week 52
Population: Analysis was performed on randomized group. Missing assessments of DAS28 were treated as no response.
Measure: Number; unit: percentage of participants
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
percentage of participants
  Week 40 | 59.2 (0.816) | 49.7 (0.822)
  Week 52 | 55.1 (1.127) | 48.3 (1.275)
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1062, Cochran-Mantel-Haenszel; DAS28 Remission Rate Difference = -9.5, 95% CI 2-sided [-20.9 to 1.8] — TCZ + PBO minus TCZ + MTX
Statistical Analysis 2: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.3611, Cochran-Mantel-Haenszel; DAS28 Remission Rate Difference = -6.8, 95% CI 2-sided [-18.2 to 4.6] — TCZ + PBO minus TCZ + MTX

7. Secondary Outcome: Percentage of Participants With DAS28 Score </=3.2 (Low DAS28)
Description: The DAS28 was derived from assessments of ESR measured in mm/h, TJC28, SJC28, and Patient's global assessment of disease activity according to 100-mm VAS. DAS28 score was calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28-ESR score could range from 0 to 10, where higher score represented higher disease activity.
Time Frame: Week 40, Week 52
Population: Analysis was performed on randomized group. Missing assessments of DAS28 were treated as no response.
Measure: Number; unit: percentage of participants
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 147 | 147
percentage of participants
  Week 40 | 76.9 (0.816) | 63.3 (0.822)
  Week 52 | 68.0 (1.127) | 62.6 (1.275)
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0228, Cochran-Mantel-Haenszel; Low DAS28 Rate Difference = -13.6, 95% CI 2-sided [-24.0 to -3.3] — TCZ + PBO minus TCZ + MTX
Statistical Analysis 2: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.3665, Cochran-Mantel-Haenszel; Low DAS28 Rate Difference = -5.4, 95% CI 2-sided [-16.3 to 5.4] — TCZ + PBO minus TCZ + MTX

8. Secondary Outcome: Change From Week 24 in Bone Erosion Score at Week 40 for Participants in the Magnetic Resonance Imaging (MRI) Substudy
Description: Bones from the wrist regions (carpal bones, distal radius, distal ulna, and metacarpal bases) and the metacarpophalangeal (MCP) joints (metacarpal heads and phalangeal bases) were assessed for erosion via MRI and scored separately based on the proportion of eroded bone compared to the 'assessed bone volume' judged from all available images. Scoring ranged from 0 (no erosion) to 10 (91-100%). Results were summed, resulting in scores from 0 to 80 for the wrist region, 0 to 150 for the MCP joints, and 0 to 230 on aggregate. A negative value for change from Week 24 in bone erosion score indicated an improvement.
Time Frame: Weeks 24, Week 40
Population: Analysis was performed on MRI subset which included all participants in the randomized group who passed MRI eligibility requirements and who had an MRI performed on or after the Week 24 visit. Here, 'Number Analyzed' signifies participants with assessment at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: Randomized Participants (TCZ + MTX) | Period 2: Randomized Participants (TCZ + PBO)
Number analyzed (Participants) | 41 | 38
units on a scale
  Week 24 | 10.66 (11.217) | 9.05 (7.926)
  Change at Week 40: number analyzed (Participants) | 39 | 33
  Change at Week 40 | -0.10 (0.844) | 0.17 (1.067)
Statistical Analysis 1: Comparison: Period 2: Randomized Participants (TCZ + MTX) vs Period 2: Randomized Participants (TCZ + PBO); ANCOVA model included Week 24 bone erosion as a covariate, treatment group, and the randomization stratification factors: DAS28 remission status at Week 24 (<2.6, >/=2.6 to </=3.2), participant anti-TNF exposure (Yes/No), baseline weight-by-dosing group (<80 kg q2w, 80-<100 kg q2w, 80-<100 kg qw, >=100 kg qw); Test type: Superiority; Estimated Mean Difference = 0.24, 95% CI 2-sided [-0.21 to 0.68], Standard Error of Mean 0.22 — TCZ + PBO minus TCZ + MTX

9. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATA) to TCZ
Description: Percentage of participants with positive results for ATA against TCZ at Baseline and at any of the post-baseline assessment time-points was reported. Participants positive at any post-baseline time points were participants who had no positivity at baseline for the same assay.
Time Frame: Baseline, Post-baseline (assessed at Weeks 12, 24, 36, 52 and at follow up [Week 60])
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. The analysis included overall study population and was not intended to compare the 2 randomized groups. 'Number Analyzed' = participants with ATA assessment at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 713
percentage of participants
  Baseline: number analyzed (Participants) | 701
  Baseline | 1.8
  Post-baseline: number analyzed (Participants) | 686
  Post-baseline | 1.5

10. Secondary Outcome: Mean TCZ Serum Concentration
Time Frame: Baseline, Weeks 12, 24, 36, 52 and follow up (Week 60)
Population: Analysis was performed on safety population. The analysis included overall study population and was not intended to compare the 2 randomized groups. 'Number Analyzed' = number of participants with assessment at specified time points.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Overall Study Population
Number analyzed (Participants) | 713
micrograms per milliliter
  Baseline: number analyzed (Participants) | 700
  Baseline | 0.01 (0.223)
  Week 12: number analyzed (Participants) | 683
  Week 12 | 8.66 (10.590)
  Week 24: number analyzed (Participants) | 641
  Week 24 | 23.38 (22.979)
  Week 36: number analyzed (Participants) | 586
  Week 36 | 25.58 (23.133)
  Week 52: number analyzed (Participants) | 66
  Week 52 | 16.46 (20.976)
  Week 60: number analyzed (Participants) | 457
  Week 60 | 6.16 (15.768)

11. Secondary Outcome: Mean Soluble Interleukin-6 (IL-6) Receptor Concentration
Time Frame: Baseline, Weeks 12, 24, 36, 52 and follow up (Week 60)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Overall Study Population
Number analyzed (Participants) | 713
nanograms per milliliter
  Baseline: number analyzed (Participants) | 695
  Baseline | 40.4 (18.14)
  Week 12: number analyzed (Participants) | 685
  Week 12 | 366.4 (179.21)
  Week 24: number analyzed (Participants) | 641
  Week 24 | 441.3 (190.78)
  Week 36: number analyzed (Participants) | 583
  Week 36 | 468.9 (211.73)
  Week 52: number analyzed (Participants) | 64
  Week 52 | 336.3 (267.20)
  Week 60: number analyzed (Participants) | 457
  Week 60 | 166.8 (211.39)

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 60
Description: Analysis was performed on safety population. The analysis included overall study population and was not intended to compare the 2 randomized groups.
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 72/713
Other Adverse Events (participants affected / at risk) | 348/713
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study Population (N=713)
Pneumonia (Infections and infestations) | 10
Cellulitis (Infections and infestations) | 3
Arthritis infective (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Abscess neck (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Encephalitis viral (Infections and infestations) | 1
Gastritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Thrombophlebitis septic (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 5
Angina unstable (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 5
Death (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study Population (N=713)
Alanine aminotransferase increased (Investigations) | 101
Hepatic enzyme increased (Investigations) | 69
Aspartate aminotransferase increased (Investigations) | 65
Liver function test increased (Investigations) | 52
Upper respiratory tract infection (Infections and infestations) | 93
Urinary tract infection (Infections and infestations) | 54
Sinusitis (Infections and infestations) | 40
Nausea (Gastrointestinal disorders) | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.